CLINICAL TRIAL: NCT01496729
Title: Single Shot Transversus Abdominis Plane (TAP) Block Versus Sham Block for Analgesia in Donors and Recipients Following Kidney Transplantation
Brief Title: Transversus Abdominis Plane (TAP) Block After Kidney Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-06622
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Transplantation, Kidney
Keywords: Kidney transplantation; Transversus abdominis plane (TAP) block
MeSH Terms: conditions — Bites and Stings | interventions — Dental Occlusion; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transversus abdominis plane (TAP) block with ropivacaine (Active Comparator): A Transversus abdominis plane (TAP) block with ropivacaine, a local anesthetic, will be performed at the end of the surgical procedure
  Interventions: Procedure: Transversus abdominis plane (TAP) block
- Sham TAP block with normal saline (Sham Comparator): A sham TAP block with normal saline will be performed at the end of the surgical procedure.
  Interventions: Procedure: Sham TAP block with normal saline

INTERVENTIONS:
Procedure: Transversus abdominis plane (TAP) block — A Transversus abdominis plane (TAP) block with ropivacaine, a local anesthetic, will be performed at the end of the surgical procedure.
  Arms: Transversus abdominis plane (TAP) block with ropivacaine
Procedure: Sham TAP block with normal saline — A sham TAP block with normal saline will be performed at the end of the surgical procedure.
  Arms: Sham TAP block with normal saline

SUMMARY:
Postoperative pain is a major problem in patients who either donate a kidney or undergo kidney transplantation. This pain is commonly treated with opioids, which can cause several side effects, ranging from pruritus, impaired vigilance, and most concerning to severe respiratory depression. This can be aggravated in the recipient by accumulation of opioid metabolites secondary to renal impairment and secretion.

Several studies have shown an opioid sparing effect of a transversus abdominis plane (TAP) block after surgery in the lower abdomen. In the proposed study, we plan to compare the impact of an ultrasound guided single shot transversus abdominis plane (TAP) block versus a ultrasound guided sham block with normal saline (placebo) on postoperative pain scores, postoperative opioid consumption, as well as patient's satisfaction.

The investigators hypothesize, that patients who receive a TAP block will have lower postoperative pain scores, lower postoperative opioid consumption as well as higher satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, English speaking, receiving a kidney transplant or donating a kidney as part of standard clinical care

Exclusion Criteria:

* Allergy to local anesthetics or opioids, coagulopathy or dementia. Patients with known history of IV drug abuse and with very high preoperative opioid requirements (defined as > 120 mg oxycodone/ day, use of methadone or fentanyl patches) will also be excluded from this study.

Coagulopathy will be assessed by the patient's history and physical. Should there be concerns regarding "easy bleeding" or "easy bruising", further workup of the patient's coagulation will be ordered (PT, PTT, INR). Since we perform the TAP block after 3-4 hours of kidney surgery, any patient with coagulopathy will most likely have been canceled prior to surgery. Therefore, we would deem any patient, who was eligible for kidney surgery, eligible for a TAP block at the end of the surgical procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pain after kidney transplantation | 24 hours
  Pain scores after kidney transplantation are measured with the visual analog scale (VAS) several times at defined times after kidney transplantation during the first 24 hours after surgery. Pain scores between the two arms of the study will be compared to each other.

SECONDARY OUTCOMES:
Use of opioids after kidney transplantation | 24 hours
  The total amount of opioids needed in the first 24 hours after kidney transplantation is recorded with the help of a patient controlled analgesia (PCA) pump and compared between the two arms of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Medical Center at Parnassus, San Francisco, California, United States